CLINICAL TRIAL: NCT02895178
Title: Lifestyle Intervention for Breast Cancer Survivors
Brief Title: Lifestyles Of Health And Sustainability for Breast Cancer Survivors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wonju Severance Christian Hospital (Other)
Responsible Party: Principal Investigator, In Deok Kong, MD, Professor, Wonju Severance Christian Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: LOHAS-BCS
Record Dates: First submitted 2016-08-21; First posted 2016-09-09 (Estimated); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Survivors; Exercise
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Exercise in breast cancer survivors (Experimental): Combined aerobic and strength exercise training for 12 weeks under supervision
  Interventions: Behavioral: Combined aerobic and strength exercise training
- No exercise in breast cancer survivors (No Intervention): Lifestyle counseling and standard of care follow up for 12 weeks
- Exercise in healthy subjects (Sham Comparator): Age-matched healthy subjects. Combined aerobic and strength exercise training for 12 weeks under supervision
  Interventions: Behavioral: Combined aerobic and strength exercise training

INTERVENTIONS:
Behavioral: Combined aerobic and strength exercise training — Subjects participate in supervised exercise sessions for 60 minutes thrice weekly and are encouraged to participate in a home-based exercise session over 30 minutes once weekly for 12 weeks.
  Arms: Exercise in breast cancer survivors; Exercise in healthy subjects

SUMMARY:
The purpose of this study is to examine the effects of exercise program on health-related physical fitness and biomarkers among breast cancer survivors.

DETAILED DESCRIPTION:
Patients and survivors of breast cancer present impaired physical fitness and various complications including acute and chronic pain, severe fatigue, limited range of motion, and bone loss attributable to anticancer treatments. Therefore, regular exercise during and following cancer treatments has been recommended to enhance physical capabilities and relieve side-effect severities, leading to an improved quality of life. Despite the known general benefits to patients with cancer, the effects of exercise on cancer-related biomarkers and their modulators remain unclear.

PRIMARY OBJECTIVES:

I. To determine whether a 12-week exercise intervention will improve components of health-related physical fitness by measuring cardiorespiratory fitness, muscular exercise capacity and flexibility in breast cancer survivors.

II. To determine whether a 12-week exercise intervention will improve risk parameters of metabolic disease by measuring changes in body composition, waist circumference, blood pressure, and circulating levels of glucose, insulin, lipids components and C-reactive protein in breast cancer survivors.

III. To determine whether a 12-week exercise intervention will conduce to changes of cancer-related biomarker by measuring in serum levels of dickkopf-related protein 1 (DKK1), secreted frizzled-related protein 1 (SFRP1), sclerostin, osteoprotegerin, osteopontin, growth differentiation factor 15 (GDF-15), insulin like growth factor 1 (IGF-1), and IGFBP-3 in breast cancer survivors.

IV. To determine whether a 12-week exercise intervention will result in a improvement in inflammatory cytokines and adipokines by measuring in serum levels of interleukin 1 beta (IL-1β), IL-10, IL-11, tumor necrosis factor alpha (TNFα), leptin and adiponectin in breast cancer survivors.

V. To determine whether a 12-week exercise intervention will conduce to changes of myokines by measuring in serum levels of brain-derived neurotrophic factor (BDNF), IL-8, IL-15, fatty acid-binding protein 3 (FABP3), leukemia inhibitory factor (LIF), follistatin, fractalkine, fibroblast growth factor 21 (FGF-21), osteonectin and irisin in breast cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Have diagnosed as a stage of I-III breast cancer
* Have undergone a lumpectomy or mastectomy
* Have completed neoadjuvant/adjuvant chemotherapy and able to initiate Exercise program
* Nonsmokers (i.e., not smoking during previous 12 months)
* Able to provide physician clearance to participate in exercise program for 12 weeks

Exclusion Criteria:

* History of chronic disease including diabetes, uncontrolled hypertension or thyroid disease
* Weight reduction >= 10% within past 6 months
* Metastatic disease
* Participate in more than 60 minutes of exercise per week in the past 6 months
* Cardiovascular, respiratory or musculoskeletal disease or joint problems that preclude moderate physical activity

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-05; Primary Completion 2023-03 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Changes of health-related physical fitness components (1). | Changes from baseline aerobic capacity at 12 weeks
  Aerobic capacity is assessed using multi-stage 20 meters shuttle run test (the maximum number of repetitions).
Changes of health-related physical fitness components (2). | Changes from baseline muscular endurance at 12 weeks
  Muscular endurance is assessed using sit-up test for 30 seconds (the maximum number of repetitions).
Changes of health-related physical fitness components (3). | Changes from baseline muscular strength at 12 weeks
  Muscular strength is assessed by the maximum voluntary strength of handgrip (kg).
Changes of health-related physical fitness components (4). | Changes from baseline muscular power at 12 weeks
  Muscular power is assessed using standing long jump test (the maximum horizontal distance of two trials, cm).
Changes of health-related physical fitness components (5). | Changes from baseline agility at 12 weeks
  Agility is assessed using 10 meters agility shuttle run test (the time taken to complete a 10 meters course is recorded, seconds).
Changes of health-related physical fitness components (6). | Changes from baseline flexibility at 12 weeks
  Flexibility is assessed using sit and reach test (the greater distance of two trials, cm)
Changes of anthropometric parameters (1). | Changes from baseline waist circumference at 12 weeks
  Waist circumference is measured at the midpoint between the lower rib margin and the iliac crest (expressed in cm).
Changes of anthropometric parameters (2). | Changes from baseline BMI at 12 weeks
  BMI calculated as body weight / height (kg per square meters).
Changes of body composition parameters (1). | Changes from baseline body fat mass at 12 weeks
  Body fat mass is measured by a bio-impedance analyzer (expressed as kg).
Changes of body composition parameters (2). | Changes from baseline lean body mass at 12 weeks
  Lean body mass is measured by a bio-impedance analyzer (expressed as kg).
Changes of body composition parameters (3). | Changes from baseline percentage body fat at 12 weeks
  Percentage body fat is calculated as body fat mass (kg) divided by weight (kg).
Changes of serum levels of Wnt signaling-related molecules (1). | Changes from baseline serum levels of DKK1 at 12 weeks
  The serum concentration of DKK1 is measured by commercial enzyme-linked immunosorbent assay kits (Minimal detectable density, 15.6 pg/ml; Standard curve range, 31.2 - 2,000 pg/ml, R&D systems).
Changes of serum levels of Wnt signaling-related molecules (2). | Changes from baseline serum levels of Sclerostin at 12 weeks
  The serum concentration of sclerostin is measured by commercial enzyme-linked immunosorbent assay kits (Minimal detectable density, 6.96 pg/ml; Standard curve range, 7.49 - 1,820 pg/ml, R&D systems).
Changes of serum levels of Wnt signaling-related molecules (3). | Changes from baseline serum levels of SFRP1 at 12 weeks
  The serum concentration of SFRP1 is measured by commercial enzyme-linked immunosorbent assay kits (Minimal detectable density, 53 pg/ml; Standard curve range, 156 - 10,000 pg/ml, USCN Life Science Inc.).
Changes of serum levels of Wnt signaling-related molecules (4). | Changes from baseline serum levels of β-catenin at 12 weeks
  The serum concentration of β-catenin is measured by commercial enzyme-linked immunosorbent assay kits (Minimal detectable density, 3.9 pg/ml; Standard curve range, 15.6 - 1000 pg/ml, Cusabio Biotech).
Changes of serum levels of Wnt signaling-related molecules (5). | Changes from baseline serum levels of WISP-1 at 12 weeks
  The serum concentration of WISP-1 is measured by commercial chemiluminescent immunoassay kits (Minimal detectable density, 0.97 pg/ml; Standard curve range, 2.74 - 2,000 pg/ml, USCN Life Science Inc.).

SECONDARY OUTCOMES:
Changes of serum levels of cancer-related molecules (1). | Changes from baseline serum levels of osteoprotegerin at 12 weeks
  The serum concentration of osteoprotegerin is measured using commercial luminex multiplexed cytokine assay panels (Minimal detectable density, 3.62 pg/ml; Standard curve range, 81.4 - 19,770 pg/ml, R&D systems).
Changes of serum levels of cancer-related molecules (2). | Changes from baseline serum levels of osteopontin at 12 weeks
  The serum concentration of osteopontin is measured using commercial luminex multiplexed cytokine assay panels (Minimal detectable density, 413 pg/ml; Standard curve range, 3.4 - 826.9 ng/ml, R&D systems).
Changes of serum levels of cancer-related molecules (3). | Changes from baseline serum levels of GDF-15 at 12 weeks
  The serum concentration of GDF-15 is measured using commercial luminex multiplexed cytokine assay panels (Minimal detectable density, 1.2 pg/ml; Standard curve range, 34 - 8,270 pg/ml, R&D systems).
Changes of serum levels of adipokines (1). | Changes from baseline serum levels of adiponectin at 12 weeks
  The serum concentration of adiponectin is measured by commercial enzyme-linked immunosorbent assay kits (Minimal detectable density, 0.891 ng/ml; Standard curve range, 3.9 - 250 ng/ml, R&D systems).
Changes of serum levels of adipokines (2). | Changes from baseline serum levels of leptin at 12 weeks
  The serum concentration of leptin is measured by commercial enzyme-linked immunosorbent assay kits (Minimal detectable density, 7.8 pg/ml; Standard curve range, 15.6 - 1,000 ng/ml, R&D systems).
Changes of serum levels of myokines (1). | Changes from baseline serum levels of BDNF at 12 weeks
  The serum concentration of BDNF is measured using commercial luminex multiplexed cytokine assay panels (Minimal detectable density, 0.32 pg/ml; Standard curve range, 10.9 - 2,650 pg/ml, R&D systems).
Changes of serum levels of myokines (2). | Changes from baseline serum levels of IL-8 at 12 weeks
  The serum concentration of IL-8 is measured using commercial luminex multiplexed cytokine assay panels (Minimal detectable density, 1.8 pg/ml; Standard curve range, 8.19 - 1,990 pg/ml, R&D systems).
Changes of serum levels of myokines (3). | Changes from baseline serum levels of IL-15 at 12 weeks
  The serum concentration of IL-15 is measured using commercial luminex multiplexed cytokine assay panels (Minimal detectable density, 1.01 pg/ml; Standard curve range, 7.7 - 18,700 pg/ml, R&D systems).
Changes of serum levels of myokines (4). | Changes from baseline serum levels of FABP3 at 12 weeks
  The serum concentration of FABP3 is measured using commercial luminex multiplexed cytokine assay panels (Minimal detectable density, 472 pg/ml; Standard curve range, 1.3 - 312.2 ng/ml, R&D systems).
Changes of serum levels of myokines (5). | Changes from baseline serum levels of LIF at 12 weeks
  The serum concentration of LIF is measured using commercial luminex multiplexed cytokine assay panels (Minimal detectable density, 9.31 pg/ml; Standard curve range, 68.1 - 16,550 pg/ml, R&D systems).
Changes of serum levels of myokines (6). | Changes from baseline serum levels of follistatin at 12 weeks
  The serum concentration of follistatin is measured using commercial luminex multiplexed cytokine assay panels (Minimal detectable density, 133 pg/ml; Standard curve range, 2.6 - 650 ng/ml, R&D systems).
Changes of serum levels of myokines (7). | Changes from baseline serum levels of fractalkine at 12 weeks
  The serum concentration of fractalkine is measured using commercial luminex multiplexed cytokine assay panels (Minimal detectable density, 64.8 pg/ml; Standard curve range, 1.3 - 325.8 ng/ml, R&D systems).
Changes of serum levels of myokines (8). | Changes from baseline serum levels of FGF-21 at 12 weeks
  The serum concentration of FGF-21 is measured using commercial luminex multiplexed cytokine assay panels (Minimal detectable density, 27 pg/ml; Standard curve range, 623 - 151,330 pg/ml, R&D systems).
Changes of serum levels of myokines (9). | Changes from baseline serum levels of SPARC (osteonectin) at 12 weeks
  The serum concentration of SPARC (osteonectin) is measured using commercial luminex multiplexed cytokine assay panels (Minimal detectable density, 97.9 pg/ml; Standard curve range, 3.4 - 829.9 ng/ml, R&D systems).
Changes of serum levels of myokines (10). | Changes from baseline serum levels of irisin at 12 weeks
  The serum concentration of irisin is measured by commercial enzyme-linked immunosorbent assay kits (Minimal detectable density, 1.29 ng/ml; Standard curve range, 0.1 - 1,000 ng/ml, Phoenix Pharmaceuticals).
Changes of serum levels of inflammatory-related cytokines (1) | Changes from baseline serum levels of IL-1 beta at 12 weeks
  The serum concentration of IL-1 beta is measured using commercial luminex multiplexed cytokine assay panels (Minimal detectable density, 0.8 pg/ml; Standard curve range, 17.8 - 4,320 pg/ml, R&D systems).
Changes of serum levels of inflammatory-related cytokines (2) | Changes from baseline serum levels of IL-10 at 12 weeks
  The serum concentration of IL-10 is measured using commercial luminex multiplexed cytokine assay panels (Minimal detectable density, 1.6 pg/ml; Standard curve range, 13.7 - 3,340 pg/ml, R&D systems).
Changes of serum levels of inflammatory-related cytokines (3) | Changes from baseline serum levels of IL-11 at 12 weeks
  The serum concentration of IL-11 is measured using commercial luminex multiplexed cytokine assay panels (Minimal detectable density, 24.7 pg/ml; Standard curve range, 0.5 - 125.4 ng/ml, R&D systems).
Changes of serum levels of inflammatory-related cytokines (4) | Changes from baseline serum levels of TNF-alpha at 12 weeks
  The serum concentration of TNF-alpha is measured using commercial luminex multiplexed cytokine assay panels (Minimal detectable density, 1.2 pg/ml; Standard curve range, 14 - 3,410 pg/ml, R&D systems).
Changes of bone mineral density | Changes from baseline bone mineral density at 12 weeks
  Bone mineral density is expressed as T-score, which is measured by a compact ultrasonometer at calcaneus (Achilles Express, GE LUNAR Corp., Madison, WI)

CONTACTS AND LOCATIONS:
Overall Officials: In Deok Kong, Professor, Study Chair — Yonsei University
Locations (1):
- Center for Exercise medicine; Yonsei University, Wŏnju, Gangwon-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim TH, Chang JS, Park KS, Park J, Kim N, Lee JI, Kong ID. Effects of exercise training on circulating levels of Dickkpof-1 and secreted frizzled-related protein-1 in breast cancer survivors: A pilot single-blind randomized controlled trial. PLoS One. 2017 Feb 8;12(2):e0171771. doi: 10.1371/journal.pone.0171771. eCollection 2017. PMID 28178355